CLINICAL TRIAL: NCT03803475
Title: Gallium-68 PSMA-11 PET Imaging in Prostate Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 185513; NCI-2019-01394 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68 labeled PSMA-11 PET PSMA (Experimental): The imaging agent (Ga-68 PSMA-11 or PSMA-HBED-CC) will be administered on an outpatient basis. It will be administered a single time intravenously prior to the PET imaging. The injected dose will be 3 to 7 millicurie (mCi) +/- 10% of 68Ga-PSMA-11.
  Interventions: Drug: Ga-68 labeled PSMA-11; Device: Positron emission tomography-computed tomography (PET/CT); Device: Positron emission tomography-magnetic resonance imaging (PET/MRI)

INTERVENTIONS:
Drug: Ga-68 labeled PSMA-11 — Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if there is presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol.
  Other Names: Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled Glu-NH-CO-NH- Lys(Ahx)-HBED- CC; Ga-68 labeled Glu-urea- Lys(Ahx)-HBED-CC; Ga-68 labeled HBED-CC PSMA
Device: Positron emission tomography-computed tomography (PET/CT) — Positron emission tomography-computed tomography (PET/CT) is a nuclear medicine technique which combines, in a single gantry, a positron emission tomography (PET) scanner and an x-ray computed tomography (CT) scanner, to acquire sequential images from both devices in the same session
  Other Names: PET-CT
Device: Positron emission tomography-magnetic resonance imaging (PET/MRI) — A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan in a single session
  Other Names: PET-MRI

SUMMARY:
The investigators are imaging patients with prostate cancer using a new Positron Emission Tomography (PET) imaging agent (Ga-68-PSMA-11) in order to evaluate its ability to detect prostate cancer.

DETAILED DESCRIPTION:
Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if there is presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol. PET imaging will begin 50-100 minutes after injection, but may be possible in certain circumstances for imaging to be delayed due to patient workflow or equipment issues

Primary Objective:

Sensitivity on a per-patient and per-region-basis (Table 1) of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy, clinical and conventional imaging follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age >= 18.
2. Histopathologically proven prostate adenocarcinoma.
3. Concern for metastatic disease in one of the following settings:

   1. Initial staging with intermediate to high risk prostate cancer.
   2. Biochemical recurrence after initial therapy.
4. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Patient unlikely to comply with study procedures, restrictions and requirements and judged by the Investigator to be unsuitable for study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ga-68 Labeled PSMA-11 PET PSMA: Participants will receive the imaging agent (Ga-68 PSMA-11 or PSMA-HBED-CC) administered in a single time intravenously prior to the Positron emission tomography (PET) imaging. The injected dose will be 3 to 7 mCi +/- 10% of 68Ga-PSMA-11.
Period: Overall Study
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Started | 485
Completed | 484
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Number analyzed (Participants) | 485
Age, Continuous [Mean (Full Range); unit: years] | 70.13 [48 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 485
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 441
  Unknown or Not Reported | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 8
  White | 408
  More than one race | 2
  Unknown or Not Reported | 38
Region of Enrollment [Number; unit: participants]
  United States | 485

OUTCOME MEASURES:

1. Primary Outcome: Detection Rate of PSMA-11 PET for Positive Disease by Prostate Specific Antigen (PSA) Group
Description: Detection rate is defined as the proportion of all patients who have prostate cancer and are true-positives confirmed by the imaging based on local reads for the detection of metastatic disease. Detection rates will be stratified based upon the PSA group at time of imaging.
Time Frame: 1 day
Population: The Number Analyzed for each Row indicates the number of participants with each detected level of PSA
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Number analyzed (Participants) | 484
proportion
  PSA Level of 0 to 0.19: number analyzed (Participants) | 29
  PSA Level of 0 to 0.19 | 0.38
  PSA Level of 0.2 to 0.49: number analyzed (Participants) | 85
  PSA Level of 0.2 to 0.49 | 0.45
  PSA Level of 0.5 to 0.99: number analyzed (Participants) | 51
  PSA Level of 0.5 to 0.99 | 0.76
  PSA Level of 1 to 1.99: number analyzed (Participants) | 49
  PSA Level of 1 to 1.99 | 0.73
  PSA Level of 2 to 4.99: number analyzed (Participants) | 107
  PSA Level of 2 to 4.99 | 0.82
  PSA Level of 5 to maximum: number analyzed (Participants) | 163
  PSA Level of 5 to maximum | 0.62

2. Primary Outcome: Detection Rate of PSMA-11 PET for Positive Disease in Prostate Bed by PSA Group
Description: Detection rate is defined as the proportion of all patients who have prostate cancer located in the prostate bed and are true-positives confirmed by the imaging based on local reads for the detection of metastatic disease. Detection rates will be stratified based upon the PSA group at time of imaging.
Time Frame: 1 day
Population: The Number Analyzed for each Row indicates the number of participants with each detected level of PSA
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Number analyzed (Participants) | 484
proportion
  PSA Level of 0 to 0.19: number analyzed (Participants) | 29
  PSA Level of 0 to 0.19 | 0.14
  PSA Level of 0.2 to 0.49: number analyzed (Participants) | 85
  PSA Level of 0.2 to 0.49 | 0.09
  PSA Level of 0.5 to 0.99: number analyzed (Participants) | 51
  PSA Level of 0.5 to 0.99 | 0.18
  PSA Level of 1 to 1.99: number analyzed (Participants) | 49
  PSA Level of 1 to 1.99 | 0.37
  PSA Level of 2 to 4.99: number analyzed (Participants) | 107
  PSA Level of 2 to 4.99 | 0.50
  PSA Level of 5 to maximum: number analyzed (Participants) | 163
  PSA Level of 5 to maximum | 0.76

3. Primary Outcome: Detection Rate of PSMA-11 PET for Positive Disease in Pelvic Nodes by PSA Group
Description: Detection rate is defined as the proportion of all patients who have prostate cancer located in the pelvic nodes and are true-positives confirmed by the imaging based on local reads for the detection of metastatic disease. Detection rates will be stratified based upon the PSA group at time of imaging.
Time Frame: 1 day
Population: The Number Analyzed for each Row indicates the number of participants with each detected level of PSA
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Number analyzed (Participants) | 484
proportion
  PSA Level of 0 to 0.19: number analyzed (Participants) | 29
  PSA Level of 0 to 0.19 | 0.10
  PSA Level of 0.2 to 0.49: number analyzed (Participants) | 85
  PSA Level of 0.2 to 0.49 | 0.27
  PSA Level of 0.5 to 0.99: number analyzed (Participants) | 51
  PSA Level of 0.5 to 0.99 | 0.51
  PSA Level of 1 to 1.99: number analyzed (Participants) | 49
  PSA Level of 1 to 1.99 | 0.24
  PSA Level of 2 to 4.99: number analyzed (Participants) | 107
  PSA Level of 2 to 4.99 | 0.34
  PSA Level of 5 to maximum: number analyzed (Participants) | 163
  PSA Level of 5 to maximum | 0.37

4. Primary Outcome: Detection Rate of PSMA-11 PET for Positive Disease in Distant Soft Tissues by PSA Group
Description: Detection rate is defined as the proportion of all patients who have prostate cancer located in the distant soft tissues and are true-positives confirmed by the imaging based on local reads for the detection of metastatic disease. Detection rates will be stratified based upon the PSA group at time of imaging.
Time Frame: 1 day
Population: The Number Analyzed for each Row indicates the number of participants with each detected level of PSA
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Number analyzed (Participants) | 484
proportion
  PSA Level of 0 to 0.19: number analyzed (Participants) | 29
  PSA Level of 0 to 0.19 | 0.10
  PSA Level of 0.2 to 0.49: number analyzed (Participants) | 85
  PSA Level of 0.2 to 0.49 | 0.09
  PSA Level of 0.5 to 0.99: number analyzed (Participants) | 51
  PSA Level of 0.5 to 0.99 | 0.10
  PSA Level of 1 to 1.99: number analyzed (Participants) | 49
  PSA Level of 1 to 1.99 | 0.18
  PSA Level of 2 to 4.99: number analyzed (Participants) | 107
  PSA Level of 2 to 4.99 | 0.30
  PSA Level of 5 to maximum: number analyzed (Participants) | 163
  PSA Level of 5 to maximum | 0.21

5. Primary Outcome: Detection Rate of PSMA-11 PET for Positive Disease in Bones (Osseous Lesions) by PSA Group
Description: Detection rate is defined as the proportion of all patients who have prostate cancer located in the bone (osseous lesions) and are true-positives confirmed by the imaging based on local reads for the detection of metastatic disease. Detection rates will be stratified based upon the PSA group at time of imaging.
Time Frame: 1 day
Population: The Number Analyzed for each Row indicates the number of participants with each detected level of PSA
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
Number analyzed (Participants) | 484
proportion
  PSA Level of 0 to 0.19: number analyzed (Participants) | 29
  PSA Level of 0 to 0.19 | 0.03
  PSA Level of 0.2 to 0.49: number analyzed (Participants) | 85
  PSA Level of 0.2 to 0.49 | 0.09
  PSA Level of 0.5 to 0.99: number analyzed (Participants) | 51
  PSA Level of 0.5 to 0.99 | 0.18
  PSA Level of 1 to 1.99: number analyzed (Participants) | 49
  PSA Level of 1 to 1.99 | 0.22
  PSA Level of 2 to 4.99: number analyzed (Participants) | 107
  PSA Level of 2 to 4.99 | 0.25
  PSA Level of 5 to maximum: number analyzed (Participants) | 163
  PSA Level of 5 to maximum | 0.26

ADVERSE EVENTS:
Time Frame: Up to 1 day
Arm/Group | Ga-68 Labeled PSMA-11 PET PSMA
All-Cause Mortality (participants affected / at risk) | 0/485
Serious Adverse Events (participants affected / at risk) | 0/485
Other Adverse Events (participants affected / at risk) | 0/485

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03803475/Prot_SAP_000.pdf